CLINICAL TRIAL: NCT02694549
Title: Prospective, Single Arm Study to Assess the Performance and Safety of CaveoVasc System for Femoral Vascular Access and Closure Device
Brief Title: CaveoVasc System - a New Femoral Vascular Access and Closure Device
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: CaveoMed GmbH (Industry)
Collaborators: MedPass International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Other
Other Study IDs: CaveoMed-2015-06
Record Dates: First submitted 2016-02-25; First posted 2016-02-29 (Estimated); Results first posted 2018-08-28 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Catheterization Via a Femoral Sheath ≤ 6Fr
Keywords: Vascular Closure Devices; Catheterization Closure Devices; Vascular Access Devices

ARMS (1):
- CaveoVasc (Experimental)
  Interventions: Device: CaveoVasc

INTERVENTIONS:
Device: CaveoVasc

SUMMARY:
The purpose of this study is to assess the performance and safety of the CaveoVasc® System for femoral vascular access and for prevention of bleeding from the femoral artery puncture site.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Patients eligible for a non-emergent diagnostic or interventional catheterization via a femoral sheath of less or equal 6Fr
* In the investigator's opinion, the patient is suitable for the CaveoVasc® System , conventional hemostasis techniques and participation in an investigational trial.
* Understand and sign the study specific written informed consent form.

Exclusion Criteria:

* Patients with significant anemia (hemoglobin <10g/DL, Hct<30).
* Patients with a baseline INR > 1.5
* Active bleeding or high bleeding risk (severe liver failure, active peptic ulcer, creatinine clearance < 30 mL/min, platelets count < 100,000 mm3), patients with chronic use of vitamin K antagonists, direct thrombin inhibitors or oral factor Xa antagonists
* Severe concomitant disease with life expectancy below 12 months
* Uncontrolled systemic hypertension
* Patients who are immunocompromised.
* Patients who need a puncture needle longer than 8 cm due to morbidity obesity
* Active systemic or cutaneous infection or inflammation
* Prior arterial surgery in abdomen and/or lower extremities
* Cardiogenic shock
* Patients who are known to be pregnant or lactating.
* Patients having a complication(s) at the femoral artery access site pre-sheath removal including hematoma, pseudoaneurysm, or arterio-venous fistula.
* Prior femoral vascular surgery or vascular graft in region of access site.
* Documented chronic peripheral arterial insufficiency preventing the use of the femoral technique
* Patients who are currently participating in another clinical trial of an investigational drug or device that has not concluded the follow-up period.
* Patients with known allergy to components of the device.
* Patients who cannot adhere to or complete the investigational protocol for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-08-09 (Actual); Primary Completion 2016-10-10 (Actual); Study Completion 2016-11-10 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- CaveoVasc: Patients treated with CaveoVasc System
Period: Overall Study
Arm/Group | CaveoVasc
Started | 12
Completed | 10
Not Completed | 2
Not completed — screen failures | 2

BASELINE CHARACTERISTICS:
Arm/Group | CaveoVasc
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Region of Enrollment [Number; unit: participants]
  Germany | 10

OUTCOME MEASURES:

1. Primary Outcome: Incidence at 30 Days After the Procedure of the Composite Endpoint of Access Site Related Major Adverse Vascular Events (MAVE).
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | CaveoVasc
Number analyzed (Participants) | 10
Participants | 2

2. Primary Outcome: Primary Performance Endpoint
Description: Device failure: Incidence at 30 days of bleedings requiring additional treatments of the puncture site
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | CaveoVasc
Number analyzed (Participants) | 10
Participants | 3

3. Secondary Outcome: Secondary Safety Endpoint
Description: Safety: Incidence of all adverse events at 30 days
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | CaveoVasc
Number analyzed (Participants) | 10
Participants | 2

ADVERSE EVENTS:
Arm/Group | CaveoVasc
Serious Adverse Events (participants affected / at risk) | 10/10
Other Adverse Events (participants affected / at risk) | 7/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CaveoVasc (N=10)
High Blood Pressure (Vascular disorders) | 1 (1)
Device deficiency : Access issue (Vascular disorders) | 3 (3)
Device Deficiency : closure issue (Vascular disorders) | 6 (6)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CaveoVasc (N=10)
Bleeding (Vascular disorders) | 2 (2)
Hematoma (Vascular disorders) | 2 (2)
Angina Pectoris (Cardiac disorders) | 1 (1)
Bleeding after procedure no compression necessary (Vascular disorders) | 1 (1)
Bleeding at the access site (Vascular disorders) | 1 (1)
Bleeding puncture site (Vascular disorders) | 1 (1)
Bleeding right groin up to 10 days after intervention (Vascular disorders) | 1 (1)
Diffuse hematoma (Vascular disorders) | 1 (1)
Hematoma and Induration right groin (Vascular disorders) | 1 (1)
Hematoma 0.9x2.3cm left groin (Vascular disorders) | 1 (1)
Hematoma right groin (Vascular disorders) | 1 (1)
High blood pressure during procedure 199/56mmHg (Cardiac disorders) | 1 (1)
not adequate placement of the device due to anatomical reason, iliac artery kinking (Vascular disorders) | 1 (1)
short confusion and loss in memory due to sedation (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes